CLINICAL TRIAL: NCT05962528
Title: Soft Contact Lens Fitting With Different Sagittal Height
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: KY2023024
Record Dates: First submitted 2023-07-16; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Type 1 group (Experimental): Toric soft lens with high sagittal height
  Interventions: Device: Soft lens
- Type 2 group (Experimental): Toric soft lens with low sagittal height
  Interventions: Device: Soft lens
- Type 3 group (Experimental): Spherical soft lens with high sagittal height
  Interventions: Device: Soft lens
- Type 4 group (Experimental): Spherical soft lens with low sagittal height
  Interventions: Device: Soft lens
- Control group (Placebo Comparator): Traditional spherical soft lens
  Interventions: Device: Soft lens

INTERVENTIONS:
Device: Soft lens — Patients were randomly fitted with five different designs of soft lenses

SUMMARY:
To evaluate whether there is a difference in subjective and objective fit of soft lenses with different sagittal height

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* No active eye disease
* 5 soft lenses for the experiment can be successfully worn and all examinations can be completed as required

Exclusion Criteria:

* Active eye disease
* BCVA less than 20/25
* Those who are too small or tight eyelids are not suitable for wearing soft lenses

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Subjective questionnaire | 1 day (Once time after wearing the soft lens)
  The subjective questionnaire is a visual quality questionnaire developed by combining previous research and clinical symptoms, including whether there is foreign body sensation, pain, dry eyes, etc.The score ranges from 0 to 4, with the higher the score, the more obvious the symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No